CLINICAL TRIAL: NCT03632278
Title: The Effectiveness of a Mindfulness Psychoeducation Program on Emotional Regulation for People With Schizophrenia: A Pilot Randomized Control Trial
Brief Title: Mindfulness Psychoeducation Program for Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: New Life Psychiatric Rehabilitation Association (Other)
Responsible Party: Principal Investigator, LAM Ho Yan, Principal investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20180531001
Record Dates: First submitted 2018-06-15; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Schizophreniform Disorders
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Participants referred to the study will be assessed at a screening examination to ensure eligibility and obtain written consent from a research assistant.
  Eligible participants will be randomly assigned to receive Mindfulness psychoeducation programme (MBPP) plus TAU or TAU.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness psychoeducation programme (Experimental): A MBPP will be conducted for 2 hours for each session, one a week for ten weeks, with 13-15 participants per group. The protocol has been developed based on the model of mindfulness-based stress reduction proposed by Kabat-Zinn (1994) and Tong et al. (2015), and the psychoeducation programmes by Chien and Lee, and Lehman and colleagues (Chien & Lee, 2010; Kabat-Zinn et al., 1992; Lehman et al., 2004; Tong et al., 2015).
  Interventions: Behavioral: Mindfulness psychoeducation Programme
- Treatment as usual (No Intervention): The usual care group will receive routine psychiatric outpatient services, including monthly psychiatric consultation and treatment by a psychiatrist, psychiatric nursing advice and brief education according to the patient's psychosocial needs. There will be community mental health services, social welfare or financial assistance supported by medical social workers, whenever necessary.
  Participants in this control may be aware that they are receiving no extra treatment which may result in negative expectancies and inflation of the treatment effect (Stoney & Johnson, 2012). To eliminate the time effect and artificially inflated intervention effect, patients in the control group will receive telephone contact once a week to discuss their disease process and daily issues.

INTERVENTIONS:
Behavioral: Mindfulness psychoeducation Programme — A MBPP will be conducted for 2 hours for each session, one a week for eight weeks. The protocol has been developed based on the model of mindfulness-based stress reduction proposed by Kabat-Zinn (1994) and Tong et al. (2015), and the psychoeducation programmes by Chien and Lee, and Lehman and colleagues (Chien & Lee, 2010; Kabat-Zinn et al., 1992; Lehman et al., 2004; Tong et al., 2015).
  The programme will be integration of mindfulness and psychoeducation to cultivate the client's mindfulness attitude. The clients will learn to apply the mindfulness in illness management and daily difficulties.
  Arms: Mindfulness psychoeducation programme

SUMMARY:
The study is the first pilot randomised controlled trial (RCT) to explore the feasibility and efficacy of Mindfulness-based psychoeducation in emotion regulation and related depressive and anxiety symptoms in people with schizophrenia.

DETAILED DESCRIPTION:
There is increasing evidence to demonstrate the safety and effectiveness of mindfulness-based psychoeducation programme (MBPP) for Chinese people with schizophrenia. A single-blind, multi-site, pragmatic randomised controlled trial conducted in Hong Kong, mainland China, and Taiwan with 300 participants consistently demonstrated significant improvement in regard to insight of illness, functioning, mental state and the length of re-hospitalisations when compared with conventional psychoeducation and Treatment As Usual (TAU) groups (Chien, 2017).

The study hypothesises that:

1. Participants receiving MBPP will decrease their use of rumination and expressive suppression, and increase the use of cognitive reappraisal compared to a control group after completion of the intervention.
2. Participants receiving MBPP attain a reduction in depressive/anxiety symptoms compared to a control group after completion of the intervention.
3. These effects are expected to be maintained through 3-month follow up with regular self-practice.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years to 65 years old
* Diagnosis with schizophrenia-spectrum disorders according to the criteria of the Diagnostic and Statistical Manual for Mental Disorders DSM-IV-TR (and the latest DSM-V) or International Classification of Diseases (ICD-10)-Classification of Mental Disorders
* Able to communicate in written and conversational Chinese/Cantonese
* Able to understand the concepts of the study and to give informed consent

Exclusion Criteria:

* Comorbid organic brain disorders or substance abuse
* Participation in any forms of cognitive therapy
* Participation and/or practice of mindfulness (in the forms of Tai Chi, Qi Gong, etc.) more than twice a week during the previous three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2018-06-03 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Emotion regulation questionnaire (ERQ) | Clients will be followed up and assessed at baseline, immediately after 8 weeks of MBI intervention (post-intervention), and 3 months post-intervention by the assessor who will be blind to participant allocation
  This is a self-report questionnaire that measures two different emotion regulation patterns: cognitive reappraisal and expressive suppression. The questionnaire has 10 items: six items reflect the reappraisal factor and four items reflect the suppressive factor. The 10 items are rated on a scale from 1 (strongly disagree) to 7 (strongly agree).

SECONDARY OUTCOMES:
Change in Short Ruminative Response Scale (SRRS) | Clients will be followed up and assessed at baseline, immediately after 8 weeks of MBI intervention (post-intervention), and 3 months post-intervention by the assessor who will be blind to participant allocation
  It comprises 10 items that are symptom-focused, self-focused, or focused on the possible causes and consequences of the depressive mood. Participants will be asked to rate on a four-point Likert scale, resulting in a possible range of scores from 22 to 88, with a higher score implying a higher level of rumination.
Change in Depression Anxiety Stress Scale (DASS-21) | Clients will be followed up and assessed at baseline, immediately after 8 weeks of MBI intervention (post-intervention), and 3 months post-intervention by the assessor who will be blind to participant allocation
  This instrument comprises three subscales including Depression, Anxiety, and Stress. The Depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest or involvement, anhedonia and inertia. The Anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic non-specific arousal. Each subscale consists of seven items. The severity ratings are made on a series of 4-point (0 to 3) scales (0 = did not apply to me at all, 3 = applied to me very much, or most of the time). The higher the subscale scores the more severe the symptoms.
Change in The Chinese version of the Psychotic Symptom Rating Scale (C-PSYRATS) | Clients will be followed up and assessed at baseline, immediately after 8 weeks of MBI intervention (post-intervention), and 3 months post-intervention by the assessor who will be blind to participant allocation
  C-PSYRATS consists of 17 items assessing the specific dimensions of hallucinations and delusions, with each item being rated on a 5-point scale from 0 (Absent) to 4 (Severe/Often/Extreme). There are two subscales including the auditory hallucinations subscale (AHS) consisting of 11 items, and the delusions subscale (DS) composed six items. The scale measures the subjective characteristics of AHS and DS including their nature, persistence, amount, distress, disruption and controllability toward the symptoms.
Change in Social and Occupational Functioning Assessment Scale (SOFAS) | Clients will be followed up and assessed at baseline, immediately after 8 weeks of MBI intervention (post-intervention), and 3 months post-intervention by the assessor who will be blind to participant allocation
  It is a single-item scale ranging from 1 to 100, with higher scores indicating higher functioning.
Change in Five Facet Mindfulness Questionnaire - Short form (FFMQ-SF) | Clients will be followed up and assessed at baseline, immediately after 8 weeks of MBI intervention (post-intervention), and 3 months post-intervention by the assessor who will be blind to participant allocation
  The FFMQ-SF is a 20-item questionnaire that measures five facets of mindfulness including observing, describing, acting with awareness, nonjudging, and non-reacting (Baer, Smith, Hopkins, Krietemeyer, & Toney, 2006). Items are scored on a 5-point scale ranging from 1 (never/very rarely true) to 5 (very often/always true). Higher scores indicate greater levels of mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Yan Lam, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- New Life Assocation, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henry JD, Rendell PG, Green MJ, McDonald S, O'Donnell M. Emotion regulation in schizophrenia: affective, social, and clinical correlates of suppression and reappraisal. J Abnorm Psychol. 2008 May;117(2):473-478. doi: 10.1037/0021-843X.117.2.473. PMID 18489225
- [Background] Aldao A, Nolen-Hoeksema S, Schweizer S. Emotion-regulation strategies across psychopathology: A meta-analytic review. Clin Psychol Rev. 2010 Mar;30(2):217-37. doi: 10.1016/j.cpr.2009.11.004. Epub 2009 Nov 20. PMID 20015584
- [Background] Chien WT, Lee IY, Wang LQ. A Chinese version of the Psychotic Symptom Rating Scales: psychometric properties in recent-onset and chronic psychosis. Neuropsychiatr Dis Treat. 2017 Mar 8;13:745-753. doi: 10.2147/NDT.S131174. eCollection 2017. PMID 28331325
- [Background] Chien WT, Thompson DR. Effects of a mindfulness-based psychoeducation programme for Chinese patients with schizophrenia: 2-year follow-up. Br J Psychiatry. 2014 Jul;205(1):52-9. doi: 10.1192/bjp.bp.113.134635. Epub 2014 May 8. PMID 24809397
- [Background] Crawford JR, Henry JD. The Depression Anxiety Stress Scales (DASS): normative data and latent structure in a large non-clinical sample. Br J Clin Psychol. 2003 Jun;42(Pt 2):111-31. doi: 10.1348/014466503321903544. PMID 12828802
- [Background] Hou J, Wong SY, Lo HH, Mak WW, Ma HS. Validation of a Chinese version of the Five Facet Mindfulness Questionnaire in Hong Kong and development of a short form. Assessment. 2014 Jun;21(3):363-71. doi: 10.1177/1073191113485121. Epub 2013 Apr 16. PMID 23596271
- [Background] Norton PJ. Depression Anxiety and Stress Scales (DASS-21): psychometric analysis across four racial groups. Anxiety Stress Coping. 2007 Sep;20(3):253-65. doi: 10.1080/10615800701309279. PMID 17999228
- [Background] O'Driscoll C, Laing J, Mason O. Cognitive emotion regulation strategies, alexithymia and dissociation in schizophrenia, a review and meta-analysis. Clin Psychol Rev. 2014 Aug;34(6):482-95. doi: 10.1016/j.cpr.2014.07.002. Epub 2014 Jul 24. PMID 25105273
- [Background] Zhang H, & Xu Y. Reliability and Validity of the Chinese Short Ruminative Responses Scale (SRRS) in Chinese Undergraduates. Psychological research(3):34-39. 2010.
- [Background] Zhao X, Zhang BR, Zhang HP, Pan L, & Zhou RL. Reliability and validity of emotion regulation questionnaire in middle school students. Chinese Journal of Clinical Psychology(1). 2015.
- [Background] Lam AHY, & Chien WT. The effectiveness of mindfulness-based intervention for people with schizophrenia: a systematic review. Neuropsychiatry (London), 6(5): 208-222. 2016.
- [Result] Chien WT, Bressington D, Yip A, Karatzias T. An international multi-site, randomized controlled trial of a mindfulness-based psychoeducation group programme for people with schizophrenia. Psychol Med. 2017 Sep;47(12):2081-2096. doi: 10.1017/S0033291717000526. Epub 2017 Apr 4. PMID 28374661